CLINICAL TRIAL: NCT06430034
Title: Contributions of 3D Photography and Stereophotogrammetry to the Evaluation of Facial Symmetrization Through Botulinum Toxin Injections, in Patients With Peripheral Facial Palsy
Brief Title: Contributions of 3D Photography and Stereophotogrammetry to the Evaluation of Facial Symmetrization by Botulinum Toxin Injections. Study of Facial Symmetry Before and After Botulinum Toxin Injections on the Face of Patients Suffering From Sequellar Peripheral Facial Paralysis
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 24IUFC01
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Peripheral Facial Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
"This is a prospective, single-center study. The main objective of our study will be to objectively evaluate the improvement of facial symmetry after botulinum toxin injection on the face in patients suffering from sequelae of peripheral facial paralysis. A secondary objective will be to assess the utility of 3D photography and stereophotogrammetry to detect and quantify facial changes relevant to this type of treatment. The number of patients included in the study is expected to be 15 at minimum. Our study will rely on 3D photographs taken with the Vectra H2 Imaging System camera device (Canfield Scientific, Inc., Fairfield, New Jersey), which will be captured before and 3 weeks to 1 month after botulinum toxin injection into the facial muscles. Various analyses of static and dynamic symmetry will be performed using the Vectra software: bi-pupillary line angle / bi-commissural line angle, superposition of healthy and pathological sides followed by RMS (root mean square) calculation, analysis of pre- and post-injection skin displacement vectors.

The results of these analyses will allow conclusions to be drawn regarding the objective efficacy of botulinum toxin injections for facial symmetrization in patients with peripheral facial paralysis, as well as to adapt injection patterns based on the severity of facial paralysis."

ELIGIBILITY:
Inclusion Criteria:

-Patients who received injections of botulinum toxin in the facial muscles, aimed at facial symmetrization at Head and Neck Institute, Nice, France at Head and Neck Institute, Nice, France.

Exclusion Criteria:

* History of corrective surgery for facial palsy, significant facial surgery, neurodegenerative diseases, the presence of skin imperfections or facial tumors that would impede a rigorous analysis of wrinkles and facial movements.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received injections of botulinum toxin in the facial muscles, aimed at facial symmetrization at Head and Neck Institute, Nice, France
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Objective assessment of facial symmetrization after botulinum toxin injection - line | Day of injection and 3-4 weeks after.
  Assessment of static and dynamic symmetry: bi-pupillary line / bi-commissural line angle - measure in degrees
Objective assessment of facial symmetrization after botulinum toxin injection | Day of injection and 3-4 weeks after.
  Assessment of static and dynamic symmetry:
  superposition of healthy and pathological sides and calculation of RMS (root mean square)
Objective assessment of facial symmetrization after botulinum toxin injection | Day of injection and 3-4 weeks after.
  Assessment of static and dynamic symmetry:
  analysis of pre- and post-injection skin displacement vectors, Before and after botulinum toxin injection.

SECONDARY OUTCOMES:
Evaluation of the importance of symmetrization based on injection patterns, types, and degrees of facial palsy. | Day of injection and 3-4 weeks after.
  Measure of symmetrization : degrees of facial palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Charles SAVOLDELLI, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU NICE, Nice, Alpes Maritimes, France